CLINICAL TRIAL: NCT03210662
Title: Phase II Study of Pembrolizumab and Fractionated External Beam Radiotherapy in Patients With Relapsed and Refractory Non-Hodgkin Lymphoma
Brief Title: Pembrolizumab and External Beam Radiation Therapy in Treating Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0341; NCI-2018-01123 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0341 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Aggressive Non-Hodgkin Lymphoma; Recurrent Mature T- Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Aggressive Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory T-Cell Non-Hodgkin Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Transformed Marginal Zone Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Non-Hodgkin | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (EBRT, pembrolizumab) (Experimental): Beginning on day 1, patients undergo fractionated EBRT daily for 5 consecutive days a week for up to 12 or 22 treatments. Patients also receive pembrolizumab IV over 1 hour on day 2. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: External Beam Radiation Therapy; Biological: Pembrolizumab

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and external beam radiation therapy work in treating patients with non-Hodgkin lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab and external beam radiation therapy may work better in treating patients with non-Hodgkin lymphoma than pembrolizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) of pembrolizumab with concurrent fractionated external beam radiotherapy (EBRT) among patients with relapsed and refractory non-Hodgkin lymphoma (NHL).

SECONDARY OBJECTIVES:

I. To determine the safety of pembrolizumab with fractionated EBRT in patients with relapsed and refractory NHL.

II. To determine the overall response rate and complete response rate (CRR) of irradiated and non-irradiated lesions to treatment with concurrent pembrolizumab and fractionated EBRT in patients with relapsed and refractory NHL.

III. To determine the progression free survival (PFS) of pembrolizumab in combination with fractionated EBRT.

IV. To determine the overall survival (OS) of pembrolizumab in combination with fractionated EBRT.

V. To determine the duration of response of irradiated and non-irradiated lesions after concurrent pembrolizumab and fractionated EBRT.

EXPLORATORY OBJECTIVES:

I. To identify tumor and peripheral blood markers predictive of response to concurrent pembrolizumab and low to moderate dose EBRT in the setting of relapsed and refractory NHL.

II. To determine if a course of hypo-fractionated EBRT can improve response after progressive disease among patients treated with fractionated EBRT and pembrolizumab.

OUTLINE:

Beginning on day 1, patients undergo fractionated EBRT daily for 5 consecutive days a week for up to 12 or 22 treatments. Patients also receive pembrolizumab intravenously (IV) over 1 hour on day 2. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one site of lymphomatous disease amenable to external beam radiation therapy (EBRT)
* Have pathologic confirmation of aggressive non-Hodgkin lymphoma (including diffuse large B cell lymphoma, transformed follicular lymphoma, transformed marginal zone lymphoma, primary mediastinal B-cell lymphoma, T cell lymphoma and NK T-cell lymphoma). Patients with indolent B cell lymphoma are excluded
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease (>= 1.5 cm in the longest diameter for nodal or extranodal disease)
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen. Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization
* Absolute neutrophil count (ANC) >= 1,000 /mcL (performed within 10 days of treatment initiation)
* Platelets >= 50,000 / mcL (performed within 10 days of treatment initiation)
* Hemoglobin >= 8 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (performed within 10 days of treatment initiation)
* Serum creatinine OR measured or calculated creatinine clearance (creatinine clearance should be calculated per institutional standard) (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 x upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (performed within 10 days of treatment initiation)
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases (performed within 10 days of treatment initiation)
* Albumin >= 2.5 mg/dL (performed within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 10 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined - contraception, for the course of the study through 120, corresponding to time needed to eliminate any Merck study treatment(s) and/or any active comparator/combination, plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Has had prior radiation therapy to the potential radiation target such that additional radiation therapy is considered unsafe by the treating radiation oncologist
* Has a history of allogeneic stem cell transplantation
* Has a diagnosis of active scleroderma or lupus or any other autoimmune disease that by the opinion of the treating radiation oncologist would put the patient at unacceptable risk of toxicity
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active Bacillus tuberculosis (TB)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study

    * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment within the past 3 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) lymphoma or lymphomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* A woman of child bearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy. Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea C Pinnix, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from MD Anderson clinics from February 2018 until October 2021
Groups:
- Total: MK-3475 at 200 mg every 21 days for 35 cycles with concurrent EBRT (unirradiated lesions)
Period: Overall Study
Arm/Group | Total
Started | 17
Completed | 0
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Total
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 59.9 [24 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Pembrolizumab With Concurrent Fractionated External Beam Radiotherapy (EBRT) Among Patients With Relapsed and Refractory Non-Hodgkin Lymphoma (NHL)
Description: Disease response will be assessed via revised Lugano classification for the response assessment of Hodgkin and non-Hodgkin lymphoma. The end of treatment assessment is determined by positron emission tomography (PET)-computed tomography (CT) imaging for patients with fluoro-deoxyglucose (FDG) avid hematologic malignancies. For patients with FDG-avid disease, the Deauville Criteria will be utilized for PET-CT scoring on a 5 point 5-point scale, in accordance with standard response criteria. A score of 1-3 is considered negative a score of 4-5 is considered positive for the presence of active lymphoma.
Time Frame: Every 3 months until withdrawal of consent, becoming lost to follow-up, or death (an average of 14 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 17
Participants | 5

2. Secondary Outcome: Progression Free Survival
Description: as for outcome 1
Time Frame: 1.8 ~ 6.5 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total
Number analyzed (Participants) | 17
Months | 2.7 [1.8 to 6.5]

3. Secondary Outcome: Overall Survival
Description: The measurement of overall survival of patients from the start of trial participation until the death of the patient.
Time Frame: Every 3 months until withdrawal of consent, becoming lost to follow-up, or death.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total
Number analyzed (Participants) | 17
Months | 6.2 [4.5 to NA] — Insufficient number of participants with events

4. Secondary Outcome: Overall and Complete Response Rate of Irradiated vs Non-Irradiated Lesions
Time Frame: Every 3 months until withdrawal of consent, becoming lost to follow-up, or death (an average of 14 months).
Measure: Number; unit: participants
Groups:
- Irradiated Lesion; Non-irradiated Lesion: MK-3475 at 200 mg every 21 days for 35 cycles with concurrent EBRT (unirradiated lesions)
Arm/Group | Irradiated Lesion | Non-irradiated Lesion
Number analyzed (Participants) | 16 | 16
participants
  PR/CR control of lesions | 10 | 3
  No PR/CR control of lesions | 6 | 13

5. Secondary Outcome: Safety of Pembrolizumab With Fractionated EBRT
Description: Assessing patients who discontinued study treatment due to toxicity/safety concerns
Time Frame: Through Study Completion (an average of 14 months)
Population: Number of Patients removed from study for Toxicity/Safety reasons
Measure: Number; unit: participants
Arm/Group | Total
Number analyzed (Participants) | 17
participants
  Participants off treatment for toxicity/safety reasons | 1
  Participants off treatment for non-safety reasons | 16

ADVERSE EVENTS:
Time Frame: Through study completion (an average of 14 months)
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 14/17
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=17)
Lung Infection (Infections and infestations) | 2 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Platelet Count Decreased (Blood and lymphatic system disorders) | 2 (2)
Hypoxia (Investigations) | 1 (1)
Delirium (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Infections and infestations) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=17)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Fatigue (General disorders) | 11 (12)
Pain (General disorders) | 3 (3)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (3)
Prutirus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypothyroidism (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 3 (4)
Lung infection (Infections and infestations) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 5 (6)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoxia (Investigations) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Malaise (General disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT03210662/Prot_SAP_002.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT03210662/ICF_001.pdf